CLINICAL TRIAL: NCT02033382
Title: Biomarkers in First Episode Schizophrenia
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 12-02903
Record Dates: First submitted 2014-01-07; First posted 2014-01-10 (Estimated); Results first posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Schizophrenia; Schizophreniform Disorder; Schizoaffective Disorder, Depressed Type
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Whole Blood
  * DNA
  * Saliva
  * Serum
  * Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Controls: Age and gender matched healthy controls
- Patients: Participants diagnosed with Schizophrenia, schizophreniform disorder, or schizoaffective disorder, depressed type that are naive to anti-psychotic treatment.

SUMMARY:
This study will identify and evaluate relevant biomarkers and structural brain imaging for understanding potential biological illness related mechanisms in medication-naïve subjects with early psychosis before and after initiation of antipsychotic medication

DETAILED DESCRIPTION:
It is currently unknown whether deterioration early in the course of psychotic illness represents medication toxicity or the natural course of the illness. The study will help clarify this issue in observing 70 schizophrenic patients before and after they are prescribed an antipsychotic via standard of care.

In addition, schizophrenia is a heterogeneous disorder and a putative brain-derived neurotrophic factor (BDNF) deficit, while possibly a common pathway, may not fully capture the biological diversity-the supplemental biomarkers will allow us to perform a more comprehensive assessment of factors contributing to clinical course. Taken together analysis of these biomarkers in relation to clinical course and in relation to healthy subjects will inform us about biological mechanisms contributing to illness onset, effects of antipsychotic medication on these mechanisms, and the predictive value of the biomarkers for clinical course. This information will provide the foundation for future early intervention trials targeting biological mechanisms utilizing a personalized medicine approach.

The baseline visit for 70 schizophrenic patients and 70 healthy age and gender matched controls consists of structural and functional MRI in addition to a blood draw for biomarkers including BDNF, inflammation markers, DNA, oxidative stress, and folate status and additionally a salivary cortisol sample collection. Biomarkers and imaging will be repeated after 8 weeks of antipsychotic treatment in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Ages 15-40 years
3. Schizophrenia, any subtype or Schizophreniform disorder
4. Sufficient proficiency in English or Spanish to complete assessments (US)

Exclusion Criteria:

1. Major depression by the Diagnostic and Statistical Manual of Mental Disorders IV criteria
2. Calgary Depression Scale for Schizophrenia (CDSS) score of 7 or greater.
3. Clinical Global Assessment of Severity of Suicidality of 3 (moderate) or greater.
4. Serious suicide attempt within three years
5. Treatment with an antipsychotic or antidepressant within the last six months
6. Active alcohol or other substance abuse or dependence within one month
7. Unstable medical illness

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will be 70 patients, ages 15-40, with first episode schizophrenia or schizophreniform disorder with onset before age 35 who are medication naive and do not meet criteria for major depression or significant suicidal ideation or substance abuse (except nicotine) and 70 age and gender matched healthy controls. Subjects will be recruited by physicians in the Bellevue Hospital emergency room, outpatient clinic and on the Bellevue psychiatric inpatient units as well as through the inpatient / outpatient services at Shanghai Mental Health Center .
  Potential subjects will be identified by clinicians and asked whether they would like to speak to a researcher. Healthy subjects will be recruited through advertising by using a flyer.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Bellevue Hospital, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Controls | Patients
Started | 83 | 82
Completed | 32 | 36
Not Completed | 51 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Patients | Total
Number analyzed (Participants) | 73 | 79 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.86 (6.40) | 25.19 (7.39) | 24.56 (6.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 33 | 39 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 73 | 74 | 147
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 0 | 2 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 73 | 79 | 152

OUTCOME MEASURES:

1. Primary Outcome: Biomarkers
Description: Compare biomarkers for inflammation, BDNF, oxidative stress, glucocorticoids and folate/methylation status in medication-naïve schizophrenia/schizophreniform subjects and matched healthy controls to identify illness-related factors.
Time Frame: Baseline
Population: Not all biomarkers were available for analysis for all subjects.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Healthy Controls | Patients
Number analyzed (Participants) | 62 | 69
pg/mL
  BDNF | 287.37 [145.99 to 722.44] | 340.83 [142.52 to 340.83]
  Thioredoxin: number analyzed (Participants) | 61 | 69
  Thioredoxin | 492.33 [324.17 to 637.67] | 420.17 [323.58 to 609.50]
  S100B: number analyzed (Participants) | 61 | 69
  S100B | 130.44 [61.14 to 265.52] | 125.13 [69.76 to 211.93]
  C-Reactive Protein: number analyzed (Participants) | 61 | 69
  C-Reactive Protein | 7610.07 [6937.90 to 9025.92] | 7631.41 [6778.62 to 9456.46]
  Interleukin 1B: number analyzed (Participants) | 61 | 69
  Interleukin 1B | 76.77 [44.41 to 225.11] | 68.82 [35.35 to 166.58]
  Interleukin 8: number analyzed (Participants) | 61 | 69
  Interleukin 8 | 63.41 [50.77 to 82.46] | 71.30 [49.79 to 83.26]
  Tumor Necrosis Factor: number analyzed (Participants) | 61 | 69
  Tumor Necrosis Factor | 92.03 [74.28 to 103.94] | 93.60 [76.02 to 105.44]
  Interferon gamma: number analyzed (Participants) | 61 | 69
  Interferon gamma | 88.96 [64.69 to 131.47] | 89.42 [70.87 to 113.86]
  Glutamate: number analyzed (Participants) | 61 | 69
  Glutamate | 105.00 [92.00 to 121.60] | 111.00 [98.20 to 128.00]
  Aspartate: number analyzed (Participants) | 61 | 69
  Aspartate | 102.32 [79.33 to 141.65] | 134.32 [86.67 to 198.31]
  Homocysteine: number analyzed (Participants) | 61 | 69
  Homocysteine | 4.79 [4.44 to 5.38] | 4.83 [4.53 to 5.26]
  Lactate: number analyzed (Participants) | 60 | 69
  Lactate | 13.28 [9.83 to 17.75] | 15.08 [11.27 to 20.34]

2. Primary Outcome: Salivary Cortisol Levels
Description: Compare biomarkers at baseline and after 8 weeks of risperidone treatment in medication-naïve schizophrenia/schizophreniform subjects to identify treatment-related factors.
  Since Blood and Saliva was only collected from First Episode participants (FEP) at week 8 (not from healthy controls) these results only report the baseline and week 8 biomarker levels for FEP participants who completed week 8.
Time Frame: Baseline and week 8
Population: Analysis was done for first episode participants who completed both Baseline and Week 8 only.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- Baseline: Biomarkers at baseline prior to risperidone treatment in medication-naïve schizophrenia/schizophreniform subjects.
- Week 8: Biomarkers at week 8 of risperidone treatment in medication-naïve schizophrenia/schizophreniform subjects.
Arm/Group | Baseline | Week 8
Number analyzed (Participants) | 29 | 29
pg/mL
  C-reactive protein | 7541.41 [6647.32 to 9445.12] | 7627.60 [6708.99 to 9474.72]
  Interleukin 1B | 68.81 [34.82 to 153.33] | 57.01 [28.18 to 168.11]
  Interleukin 8 | 74.34 [50.02 to 93.98] | 65.79 [51.16 to 82.38]
  Interferon gamma | 95.26 [73.44 to 117.90] | 98.14 [61.71 to 124.71]
  Tumor necrosis factor | 93.60 [75.75 to 107.69] | 89.45 [71.25 to 109.15]
  Aspartate | 3.71 [2.60 to 4.55] | 4.75 [3.76 to 6.37]
  Glutamate | 5.21 [4.54 to 6.20] | 5.29 [4.77 to 6.33]
  Lactate | 4.49 [3.11 to 5.21] | 3.95 [2.75 to 6.11]
  Homocysteine | 4.78 [4.51 to 5.11] | 5.02 [4.75 to 5.31]
  BDNF | 465.98 [145.23 to 1965.72] | 356.20 [218.79 to 1040.88]
  Thioredoxin | 417.50 [291.67 to 547.75] | 405.33 [326.92 to 519.25]
  S100B | 154.63 [91.25 to 299.88] | 111.39 [49.78 to 278.73]

3. Primary Outcome: Salivary Cortisol Levels
Description: Compare biomarkers for stress (salivary cortisol) in medication-naïve schizophrenia/schizophreniform subjects and matched healthy controls to identify illness-related factors.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: µg/dL
Arm/Group | Healthy Controls | Patients
Number analyzed (Participants) | 54 | 46
µg/dL | 4.88 [3.19 to 7.51] | 6.56 [4.18 to 8.98]

4. Primary Outcome: Change in Salivary Cortisol Levels
Description: Compare salivary cortisol at baseline and after 8 weeks of risperidone treatment in medication-naïve schizophrenia/schizophreniform subjects to identify treatment-related factors.
  Since Blood and Saliva was only collected from First Episode participants (FEP) at week 8 (not from healthy controls) these results only report the baseline and week 8 biomarker levels for FEP participants who completed week 8.
Time Frame: Baseline and week 8
Population: Analysis was done for first episode subjects who completed both Baseline and Week 8 only.
Measure: Median (Inter-Quartile Range); unit: µg/dL
Groups:
- Baseline: salivary cortisol at baseline prior to risperidone treatment in medication-naïve schizophrenia/schizophreniform subjects.
- Week 8: salivary cortisol at week 8 of risperidone treatment in medication-naïve schizophrenia/schizophreniform subjects.
Arm/Group | Baseline | Week 8
Number analyzed (Participants) | 19 | 19
µg/dL | 7.41 [1.89 to 9.17] | 4.36 [2.37 to 8.20]

5. Secondary Outcome: Left Hippocampal Volumetric Integrity (HVI)
Description: Compare hippocampal volume in medication-naïve schizophrenia/schizophreniform subjects and healthy controls and examine whether biomarkers predict differences between groups in baseline hippocampal volume.
Time Frame: Baseline
Measure: Median (Inter-Quartile Range); unit: % of hippocampal volumetric integrity
Arm/Group | Healthy Controls | Patients
Number analyzed (Participants) | 54 | 57
% of hippocampal volumetric integrity | .9512 [.8501 to .9825] | .9275 [.8256 to .9689]

6. Secondary Outcome: Cognitive Performance
Description: Compare cognitive performance on the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB) in medication- naïve schizophrenia/schizophreniform subjects and healthy controls and examine whether biomarkers predict differences between groups in baseline cognitive performance. The composite score on the MCCB is calculated by the software using all tests administered. The composite score is a t-score assuming the mean score (50%) is the normative performance of the general population. The composite score ranges from 0-100 with a standard deviation of 10. A score greater than 50 implies a score better than the average population norm and a score less than 50 indicates performance worse than the general population norm.
  For schizophrenia subjects who complete 8 weeks of antipsychotic treatment, week 8 MATRICS testing results will be used to minimize the effect of psychosis on cognitive performance.
Time Frame: Baseline, week 8
Population: Data provided only for subjects who completed assessments at both time points.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Healthy Controls | Patients
Number analyzed (Participants) | 36 | 30
units on a scale
  Baseline MCCB Composite Score | 47.50 [41 to 53] | 34 [24.5 to 45.25]
  Week 8 MCCB Composite Score | 49.50 [44.25 to 54] | 42.50 [32.25 to 49]

7. Secondary Outcome: Annualized Change in Left Hippocampal Volume Integrity
Description: Compare hippocampal volume in medication-naïve schizophrenia/schizophreniform subjects before and after 8 weeks treatment with antipsychotic to assess evidence for early neurotoxicity.
  This outcome measure reports annualized rate of change in Left Hippocampal Volume Integrity (LHVI) because a few participants had a delay in their week 8 visit.
Time Frame: Baseline, week 8
Population: This analysis includes participants that completed both baseline and week 8 visits.
Measure: Median (Inter-Quartile Range); unit: Percentage of standard hippocampal vol.
Arm/Group | Healthy Controls | Patients
Number analyzed (Participants) | 31 | 24
Percentage of standard hippocampal vol. | 0.004535 [-0.0151 to 0.0350] | -0.03027 [-0.0817 to 0.00004]

ADVERSE EVENTS:
Arm/Group | Healthy Controls | Patients
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/79
Other Adverse Events (participants affected / at risk) | 0/73 | 1/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy Controls (N=73) | Patients (N=79)
Blurred Vision (Eye disorders) | 0 (0) | 1 (1) — Patient reported blurred vision
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) — BP sitting 130/100, standing 130/95

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No